CLINICAL TRIAL: NCT07390552
Title: A Prospective, Randomized, Double-blinded, Placebo-controlled, 4-Parallel Arm, Multi-center, Phase 2 Trial to Evaluate Efficacy and Safety of Orally Administered PLH-2301 in Elderly Patients With Sarcopenia
Brief Title: A Study of PLH-2301 in Subjects With Sarcopenia
Acronym: PLH-2301_P2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pluto Inc. (Industry)
Collaborators: Symyoo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLH-2301_P2
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sarcopenia in Elderly
Keywords: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects receive placebo orally in the morning, afternoon, and evening for 12 weeks.
  Interventions: Drug: Placebo
- PLH-2301 200mg (Experimental): Subjects receive PLH-2301 in the morning and placebo in the afternoon and evening for 12 weeks.
  Interventions: Drug: PLH-2301; Drug: Placebo
- PLH-2301 400mg (Experimental): Subjects receive PLH-2301 in the morning and evening and placebo in the afternoon for 12 weeks.
  Interventions: Drug: PLH-2301; Drug: Placebo
- PLH-2301 600mg (Experimental): Subjects receive PLH-2301 in the morning, afternoon, and evening for 12 weeks.
  Interventions: Drug: PLH-2301

INTERVENTIONS:
Drug: PLH-2301 — PLH-2301 administered orally according to assigned dosing regimen.
  Arms: PLH-2301 200mg; PLH-2301 400mg; PLH-2301 600mg
Drug: Placebo — Matching placebo administered orally according to assigned dosing regimen.
  Arms: PLH-2301 200mg; PLH-2301 400mg; Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of PLH-2301 in subjects with sarcopenia.

Eligible subjects aged 65 years and older will be randomized to receive placebo or one of three dose levels of PLH-2301 once daily for 12 weeks.

The primary objective is to assess the effect of PLH-2301 on physical function compared with placebo.

DETAILED DESCRIPTION:
Sarcopenia is a progressive and generalized skeletal muscle disorder associated with loss of muscle strength, physical performance, and quality of life in older adults. Currently, there are limited approved pharmacological treatment options for sarcopenia.

This Phase 2 study is designed to evaluate the efficacy and safety of PLH-2301 in subjects with sarcopenia. Approximately 168 eligible subjects will be randomized in a 1:1:1:1 ratio to receive placebo or PLH-2301 at dose levels of 200 mg, 400 mg, or 600 mg administered orally once daily for 12 weeks.

The primary efficacy endpoint is the change from baseline in the Short Physical Performance Battery (SPPB) total score at Week 12. Secondary endpoints include changes in gait speed, chair stand performance, handgrip strength, appendicular skeletal muscle mass, and health-related quality of life. Safety will be assessed throughout the study by monitoring adverse events, laboratory tests, vital signs, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 65 years or older at the time of consent
* Diagnosis of sarcopenia based on predefined diagnostic criteria
* Short Physical Performance Battery (SPPB) total score within the protocol-defined range at screening
* Stable body weight for at least 3 months prior to screening
* Able to walk independently with or without assistive devices
* Willing and able to comply with study procedures
* Provided written informed consent prior to any study-specific procedures

Exclusion Criteria:

* History of clinically significant neuromuscular or musculoskeletal disorders that could affect muscle function
* Uncontrolled cardiovascular, hepatic, renal, or metabolic disease
* Use of medications known to affect muscle mass or function within the protocol-defined washout period
* Participation in another interventional clinical trial within 3 months prior to screening
* Any medical or psychiatric condition that, in the investigator's opinion, would interfere with study participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Short Physical Performance Battery (SPPB) total score | Baseline to Week 12
  Change from baseline in the Short Physical Performance Battery (SPPB) total score.
  The Short Physical Performance Battery is a composite measure of lower extremity function with total scores ranging from 0 to 12, where higher scores indicate better physical performance.

SECONDARY OUTCOMES:
Change from baseline in gait speed | Baseline to Week 12
  Change from baseline in chair stand test time as a component of physical performance
Change from baseline in chair stand test time | Baseline to Week 12
  Change from baseline in chair stand test time as a component of physical performance
Change from baseline in handgrip strength | Baseline to Week 12
  Change from baseline in handgrip strength measured using a dynamometer
Change from baseline in appendicular skeletal muscle mass | Baseline to Week 12
  Change from baseline in appendicular skeletal muscle mass measured by bioelectrical impedance analysis
Change from baseline in Sarcopenia Quality of Life (SarQoL-K) total score | Baseline to Week 12
  Change from baseline in the Sarcopenia Quality of Life questionnaire (SarQoL-K) total score.
  The SarQoL-K total score ranges from 0 to 100, with higher scores indicating better quality of life.

OTHER OUTCOMES:
Treatment compliance rate | Throughout the 12-week treatment period
  Compliance with study medication, dietary intervention, and exercise program was monitored throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Ahe Lee, Study Director — Pluto Inc.
Locations (3):
- South Korea (3):
  - Korea University Anam Hospital, Seoul, Seoul
  - Seoul St. Mary's Hospital, Seoul, Seoul
  - Korea University Guro Hospital, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No